CLINICAL TRIAL: NCT00266500
Title: Body Heat Content and Dissipation in Obese and Normal Weight Adults
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060038; 06-CH-0038
Record Dates: First submitted 2005-12-16; First posted 2005-12-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-10-28

CONDITIONS: Obesity
Keywords: Adipose Tissue; Weight Gain; Overweight; Thermogenesis; Deep Body Temperature; Adult; Exercise
MeSH Terms: conditions — Obesity; Weight Gain; Overweight; Motor Activity

SUMMARY:
This study will investigate how different parts of the body lose body heat and will measure the heat released by specific areas such as the limbs and abdomen. Animal studies suggest that dissipation of body heat may affect energy expenditure, and therefore, body weight. This study will explore the relationship between obesity and heat in humans.

Healthy people 18 years of age and older who are of normal weight or who are obese and who are not taking medications for obesity-related medical conditions may be eligible for this study. Candidates must have a body mass index (BMI) between 18 and 25 kg/m2 for normal weight subjects or a BMI greater than 30 kg/m2 for obese subjects. All candidates must weigh less than 300 pounds. Women must have a normal menstrual cycle or be postmenopausal.

Participants undergo the following procedures in a single day on an outpatient basis:

* Medical history, physical examination, blood and urine tests and electrocardiogram.
* DEXA and MRI scans of the trunk and limbs to measure the amounts of muscle, bone and fat in the body. For the DEXA scan, the subject lies on a table while a very small dose of x-rays is passed through the body. For the MRI, the subject lies on a table that is moved into a steel cylinder. A magnetic field and radio waves produce images that are used to measure fat in the trunk of the body, thighs, and arms.
* Infrared photography of hands, front of thigh, and abdomen. A special camera is used to measure the heat leaving the body.
* Bicycle exercise test. The subject exercises on a stationary bicycle while the heart rate, heart rhythm, blood pressure and oxygen consumption are measured. The pedal resistance is increased gradually until the subject can no longer exercise and then the resistance is gradually decreased for cool-down.

Participants who qualify for the second part of the study undergo the following procedures during a 5-day in-hospital stay:

* Temperature measurements. Body temperature is measured in the ear canal. Skin temperature is measured with small round adhesive temperature-sensing patches placed on the abdomen and limbs for up to 5 days.
* Measurement of body radiowaves. A remote sensing device is used to measure microwaves that are naturally released from the body.
* Infrared photography of hands, front of thigh and abdomen is done several times during the study.
* Application of mild coolness to hands, thigh and abdomen. The subject's hand is exposed to mild coolness first by immersion in cool water, then by a cool-water spray, then by a cooled pad placed on the hand, and finally, with a device applied to the hand that cools and has a gentle vacuum. The abdomen and thigh are similarly exposed. During each test, an infrared camera records how heat is released by the body.
* Temperature effects of a "meal." The subject drinks lemon-flavored sugar water to measure the body's response.
* Bicycle exercise test. The subject exercises on three different occasions. During or after some of the tests, mild cooling is applied to the abdomen, front of the thigh, or hands.
* Measurement of exhaled air (indirect calorimetry). The subject wears a hood that collects and analyzes exhaled air for 15- to 30-minute periods.
* Photography and videotaping. The subject is photographed and videotaped. The images do not include views of any private parts, and the subject's identity is protected.

DETAILED DESCRIPTION:
Animal models suggest that dissipation of body heat is an important physiological process that may affect energy expenditure, and thus may possibly modulate body weight. It is unknown, however, if deficient dissipation of heat can contribute to human obesity, or if obesity induces deficits in heat dissipation, and the relationship between obesity and heat in humans is largely unexplored.

We propose to study obese (BMI greater than or equal to 30 kg/m(2)) and normal weight (BMI less than or equal to 25 kg/m(2)) adults to determine possible obesity-related differences in: 1) regional body temperature heterogeneity (i.e., presence of localized areas of heat retention), 2) the extent to which locally retained heat may be co-localized with deep fat depots, 3) the effectiveness of specific body loci (e.g., the distal extremities) as dissipaters of heat, and 4) the ability of approaches that alter heat dissipation to modify deep-body temperature heterogeneity.

It is hoped that the results of this study will provide preliminary evidence for future studies that attempt to facilitate weight loss in obese subjects through effective, guided applications of heat management.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify if they meet the following criteria:

1. Good general health. Individuals taking medications for obesity-related co-morbid conditions will generally be excluded, but will be considered on a case-by-case basis. Participants will be nonsmokers.
2. Age greater than or equal to 18 years.
3. Body Mass Index (BMI) between 18 and 27 kg/m(2) for normal weight subjects or BMI greater than or equal to 30 kg/m(2). To maximize differences between groups, overweight but not obese adults will not be studied. Body weight will be less than 300 pounds (136 kg), however, because DXA scanners at the Clinical Center cannot scan individuals of greater size).
4. For women with childbearing potential, a negative pregnancy test at the initial evaluation. Since these subjects have to undergo an X-ray screening, for safety purposes pregnant women will be excluded from participation in the study.
5. For women, a normal menstrual cycle or post menopausal status. Women with normal cycles will be studied between 1-3 weeks following their last menstrual period.

EXCLUSION CRITERIA (Overweight Subjects):

Volunteers will be excluded (and referred to treatment as needed) for the following reasons:

1. Presence of major illnesses: renal (serum creatinine greater than 1.6), hepatic (AST/ALT greater than 3 times upper limit of normal range used in Clinical Center assays), gastrointestinal, most endocrinologic (e.g., Cushing syndrome, hyper- or untreated hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication or sleep-apnea related disorders). The presence of the 'hunting' reflex will not exclude patients.
2. Pregnancy.
3. Individuals who have a current substance abuse, including smoking, or a psychiatric disorder or other condition that in the opinion of the investigators would impede competence or compliance, or possibly hinder completion of the study;
4. Subjects who regularly use prescription medications. Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting the study. Individuals taking medications for most conditions will be excluded, but medication use will be considered on a case-by-case basis.
5. Weight change of more than 3% of body weight in the past two months.
6. Areas to be visualized by IR are deemed by the investigators to be too hirsute to allow accurate measurement of underlying tissues.
7. Fat depth in areas to be measured is more than 4 cm.
8. Long nails that would preclude wearing snug-fitting surgical gloves.
9. Weight in excess of 300 lbs (136 kg) that would preclude being scanned by Clinical Center DXA machines.
10. Individuals that regularly participate in high-intensity physical activity, as determined by either self-report or analysis of the Past Year Total Physical Activity Questionnaire (PYTPAQ)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-12-12; Study Completion 2014-10-28

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Finkelstein EA, Ruhm CJ, Kosa KM. Economic causes and consequences of obesity. Annu Rev Public Health. 2005;26:239-57. doi: 10.1146/annurev.publhealth.26.021304.144628. PMID 15760288
- [Derived] Heikens MJ, Gorbach AM, Eden HS, Savastano DM, Chen KY, Skarulis MC, Yanovski JA. Core body temperature in obesity. Am J Clin Nutr. 2011 May;93(5):963-7. doi: 10.3945/ajcn.110.006270. Epub 2011 Mar 2. PMID 21367952
- [Derived] Savastano DM, Gorbach AM, Eden HS, Brady SM, Reynolds JC, Yanovski JA. Adiposity and human regional body temperature. Am J Clin Nutr. 2009 Nov;90(5):1124-31. doi: 10.3945/ajcn.2009.27567. Epub 2009 Sep 9. PMID 19740972